CLINICAL TRIAL: NCT01837238
Title: Efficacy of Beta-Hydroxy-Beta-Methylbutyrate (HMB) Supplementation in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Renal Reserach Institute
Record Dates: First submitted 2013-02-01; First posted 2013-04-23 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Complication of Dialysis; Chronic Kidney Disease; Muscle Loss; End Stage Renal Disease
Keywords: hemodialysis; physical function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Muscular Atrophy; Kidney Failure, Chronic | interventions — beta-hydroxyisovaleric acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- beta-hydroxy beta-methylbutyrate (Experimental): Calcium-HMB (3g) will be consumed daily for 6 months by all participants assigned to the HMB group.
  Interventions: Dietary Supplement: HMB
- Placebo (Placebo Comparator): The placebo group will consume non-nutritive placebo pills daily for 6 months.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: HMB — Following this initial round of testing,participant will be assigned to daily HMB supplementation for 6 months. You will be asked to consume a 1000mg HMB capsule 3 times per day, 7 days per week, for 6 months.
  Other Names: beta-hydroxy-beta-methylbutyrate, calcium-hmb
  Arms: beta-hydroxy beta-methylbutyrate
Dietary Supplement: placebo — The placebo group will consume non-nutritive placebo pills daily for 6 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of 6 months of daily beta-hydroxy beta-methylbutyrate (HMB) supplementation on the physical function and the health of bones, arteries and heart in hemodialysis patients.

DETAILED DESCRIPTION:
Patients with renal failure receiving hemodialysis experience an increased rate of skeletal muscle protein catabolism which is associated with a number of co-morbid conditions including declines in muscle mass and strength, significantly increased fall risk, and reduced quality of life (QOL. Therefore, interventions to prevent muscle loss in hemodialysis are needed. Pharmacological agents have been investigated to treat muscle loss in dialysis patients; however, many of these treatments are expensive and have undesirable side effects. As a result, low-cost interventions designed to attenuate losses in muscle mass and strength in hemodialysis patients are needed.

Beta-hydroxy beta-methylbutyrate (HMB) represents a potential low-cost nutritional intervention to attenuate muscle loss in hemodialysis patients. HMB is a metabolite of the amino acid leucine that has been shown to safely increase muscle mass in other clinical populations with prevalent muscle loss, such as the elderly, cancer, and AIDS patients primarily through reductions in skeletal muscle protein catabolism. The primary purpose of the trial is to determine if oral supplementation with HMB attenuates muscle loss, improves muscle strength, physical function, fall risk and QOL in hemodialysis patients. Alterations in protein and gene expression associated with skeletal muscle protein turnover will be measured to investigate the mechanism for changes in our primary outcomes. We hypothesize that HMB supplementation will attenuate declines in muscle size and strength in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Must be receiving hemodialysis treatment.
* Must be willing to be randomized to HMB or placebo for 6 months
* Must receive physician clearance to participate

Exclusion Criteria:

* Bodyweight > 350 lbs
* Currently taking an HMB supplement or HMB containing products (eg. Ensure)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in lean mass over 6 months | 6 months
  Lean mass will be assessed via DXA at baseline and after 6 months of HMB supplementation.

SECONDARY OUTCOMES:
Change in physical function over 6 months | 6 months
  Physical function will be assessed via isokinetic dynamometry and shuttle walk test at baseline and after 6 months of HMB supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wilund, PhD, Principal Investigator — Kinesiology & Community Health, UIUC
Locations (1):
- University of Illinois, Urbana, Illinois, United States